CLINICAL TRIAL: NCT05019222
Title: Comparison of Quality of Recovery (QoR)-15 Scores According to the Use of Anesthetics During General Anesthesia in the Cervical Spine Surgery Patients: Sevoflurane vs. Remimazolam
Brief Title: Comparison of Postoperative QoR-15 Scores Between Sevoflurane and Remimazolam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Myoung Hwa Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3-2021- 0257
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Anterior Cervical Discectomy and Fusion (ACDF) Surgery
Keywords: Cervical surgery; Quality of Recovery; Remimazolam; sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1) Sevoflurane group (Experimental): Sevoflurane based inhalation anesthesia
  Interventions: Drug: Sevoflurane based inhalation anesthesia
- Arm 2) Remimazolam group (Active Comparator): Remimazolam based total intravenous anesthesia
  Interventions: Drug: Remimazolam based total intravenous anesthesia

INTERVENTIONS:
Drug: Sevoflurane based inhalation anesthesia — Sevoflurane group will be inducted with bolus of propofol 1% and maintained with sevofulrane as inhalation and TCI Minto model of remifentanil for general anesthesia.
  Arms: Arm 1) Sevoflurane group
Drug: Remimazolam based total intravenous anesthesia — Remimazolam group will be inducted with remiamazolam at 6 mg/kg/h and maintained with remimazolam at 0.5-1.5 mg/kg/h and TCI Minto model of remifentanil for general anesthesia.
  Arms: Arm 2) Remimazolam group

SUMMARY:
The purpose of the study is to compare the quality of recovery (QoR)-15 scores according to the use of maintenance anesthetics in the cervical spine surgery. Total intravenous anesthesia (TIVA) have been known to help reducing risks of postoperative nausea/vomiting and malignant hyperthermia. However, it is still not enough to explain which is better between TIVA or inhalation anesthesia. In particular, there is no study to investigate overall postoperative functional recovery via QoR-15 in patients receiving TIVA with remimazolam. The hypothesis of the investigators study is that, in patients with cervical spine surgery, total intravenous anesthesia based on remimazolam can improve the the quality of recovery compared to inhalation anesthesia based on sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who aged 20-70 years
* ASA-PS: 1-3
* BMI < 30
* Anterior cervical discectomy and fusion surgery

Exclusion Criteria:

* Tolerance or hypersensitivity to benzodiazepine
* Dependence or addiction to psychotropic drugs or alcohol
* Pregnant women, subjects who lack the ability to make decisions and susceptible to voluntary participation decisions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
The difference between two groups (sevoflurane vs. remimazolam) in QoR-15 scores | postoperative day 1
  The difference of scores in the Quality of Recovery (QoR)-15 survey on POD 1 Total 0-150, 0 (minimum), 150 (maximum), Higher scores means better.

CONTACTS AND LOCATIONS:
Locations (1):
- Myung Hwa Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No